CLINICAL TRIAL: NCT00398541
Title: Evaluation of the Antihypertensive Effect of Hyzaar(R) and Cognitive Function of Hypertensive Patients
Brief Title: Evaluation of the Antihypertensive Effect of Hyzaar(R) and Cognitive Function of Hypertensive Patients (0954A-322)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-322; MK0954A-322; 2006_048
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination

INTERVENTIONS:
Drug: losartan potassium (+) hydrochlorothiazide — losartan potassium (+) hydrochlorothiazide combination will be titrated upwards according to the following scheme: losartan potassium 50/hydrochlorothiazide 12.5 then losartan potassium 100/hydrochlorothiazide 12.5 then losartan potassium 100/hydrochlorothiazide 25
  Other Names: MK954A; Hyzaar

SUMMARY:
Evaluate the antihypertensive and neuroprotective effects of Hyzaar(R) in elderly subjects in comparison with Natrilix(TM).

ELIGIBILITY:
Inclusion Criteria:

* ACEi or ARB naive or not taking ACEi or ARB concurrently for at least one month before the run-in period
* Be able to carry out his or her own daily activity
* - Be at least 50 years old at inclusion in the study Be diagnosed with mild to moderate hypertension, treated or untreated
* Literate
* Not taking any cognitive-enhanced agent at baseline
* Present with a memory complain ( spontaneous or informed by caregiver)

Exclusion Criteria:

* Congestive heart failure with NYHA class >2
* Renal failure or renal insufficiency with serum creatinine >1.4mg/dl
* chronic severe liver disease with abnormal GPT and GOT >2 times of upper normal limits
* Diagnosed with major depression when entering the study
* Foreign language as his or her mother tongue so that the test results will not be reliable
* History of stroke or transient ischemic attack (stroke is defined as focal neurological sign progressing stepwise)
* Hypersensitive to the active ingredient and any other component of losartan potassium and indapamide tablets
* Major hearing loss/deafness and/or major visual impairment/blindness preventing from performing the tests
* Myocardial infarction within the past 6 months
* Single functioning kidney
* Anuria

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2007-04-10 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychological tests and blood pressure after treatment of 12 weeks | after treatment of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC